CLINICAL TRIAL: NCT00777465
Title: Prognostic Value of Acute Kidney Injury After Cardiac Surgery According to Kidney Disease: Improving Global Outcomes Definition and Staging (KDIGO) Criteria
Brief Title: Acute Kidney Injury After Cardiac Surgery Based on KDIGO Criteria
Status: Completed | Type: Observational
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Mauricio de Nassau Machado, Cardiologist in-chief - Coronary Care Unit, Hospital de Base
Other Study IDs: CAAE-3436.0.000.140-08
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Kidney failure; Risk factors; Clinical outcomes; Cardiac valve surgery; Coronary artery bypass grafting; Morbidity; Mortality
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- KDIGO 0: Patients with no acute kidney injury after cardiac surgery
- KDIGO 1: Patients with acute kidney injury KDIGO stage 1 after cardiac surgery (Increase in SCr by ≥ 0.3 mg/dL (≥ 26.5 lmol/L) or 1.5 to 1.9 times baseline)
- KDIGO 2: Patients with acute kidney injury KDIGO stage 2 after cardiac surgery (2.0 to 2.9 times baseline SCr)
- KDIGO 3: Patients with acute kidney injury KDIGO stage 3 after cardiac surgery (3.0 times baseline or more; or increase in SCr to ≥ 4.0 mg/dL; or initiation of renal replacement therapy)

SUMMARY:
The aim of this study was to apply the acute kidney injury criteria based on KDIGO classification in a population of patients undergoing cardiac surgery [coronary artery bypass grafting (CABG) or cardiac valve surgery (CVS)] and evaluate its impact as a predictor of 30-day mortality.

DETAILED DESCRIPTION:
This was a single center study. We evaluated retrospectively patients from the Cardiac Surgery Intensive Care Unit in Hospital de Base, São José do Rio Preto Medical School, São Paulo, Brazil. Demographics, type of surgery, laboratory data and preoperative, perioperative, and postoperative information were retrieved from a prospectively collected database of 2878 patients older than 18 years undergoing isolated CABG (1786) or CVS (1092), from January 2003 to June 2013. After applying the exclusion criteria (51 patients with incomplete data and 23 patients with end-stage kidney disease) we analyzed 2804 patients in total, 1738 (62%) underwent CABG and 1066 (38%) underwent CVS.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing isolated coronary artery bypass grafting or cardiac valve surgery.

Exclusion Criteria:

patients with incomplete data and patients with end-stage kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected consecutively after cardiac surgery (CABG or CVS) in a setting of postoperative intensive care unit.
Sampling Method: Probability Sample
Enrollment: 2804 (Actual)
Dates: Start 2003-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury after cardiac surgery as a independent predictor of 30-day mortality | 30 days
  To test the hypothesis that the acute kidney injury based on KDIGO criteria after cardiac surgery is a independent predictor of 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Lilia N Maia, PhD, Study Director — São José do Rio Preto Medical School
Locations (1):
- Hospital de Base, São José do Rio Preto, São Paulo, Brazil